CLINICAL TRIAL: NCT06453850
Title: Safety and Performance Evaluation of a New Catheter Range for Lead Implantation At Interventricular Septum
Acronym: POLARIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DARI01 - POLARIS
Record Dates: First submitted 2024-05-29; First posted 2024-06-12 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Bradycardia; Cardiac Resynchronization Therapy; Left Bundle Branch Area Pacing
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- FLEXIGO delivery catheter (Experimental)
  Interventions: Device: Use of FLEXIGO delivery catheter

INTERVENTIONS:
Device: Use of FLEXIGO delivery catheter — Use of FLEXIGO delivery catheter for implantation of ventricular pacing lead

SUMMARY:
The purpose of the clinical investigation is to evaluate the safety of the FLEXIGO delivery catheter for transvenous pacing lead implantation.

ELIGIBILITY:
Inclusion criteria (phase I):

* Patient indicated for cardiac pacing according to the most recent guidelines from the European Society of Cardiology (ESC)
* Patient planned for a de novo implantation of any Single Chamber (SR) or Dual Chamber (DR) CE marked pacemaker
* Patient planned for a catheter-guided implantation in the interventricular septum area
* Patient planned for the implantation of any CE marked ventricular pacing lead compatible with the FLEXIGO delivery catheter
* Patient reviewed, signed and dated the Informed Consent Form (ICF)

Inclusion criteria (phase II):

* Patient indicated for cardiac pacing or CRT according to the most recent guidelines from the ESC
* Patient planned for a de novo implantation of any SR or DR CE marked pacemaker, or any CE marked CRT-D
* Patient planned for a catheter-guided implantation in the interventricular septum area
* Patient planned for the implantation of any CE marked ventricular pacing lead compatible with the FLEXIGO delivery catheter
* Patient reviewed, signed and dated the ICF

Exclusion criteria (phase I):

* Patient planned for a device upgrade, or a device or a lead replacement
* Patient with a congenital heart disease
* Patient with significant hypertrophic cardiomyopathy, cardiac amyloidosis or obstructive hypertrophic cardiomyopathy
* Patient with a Left Ventricular Ejection Fraction (LVEF) ≤ 35%
* Patient already enrolled in another clinical investigation that could confound the results of this clinical investigation (e.g., clinical investigations involving intra-cardiac device)
* Patient implanted despite a contraindication for cardiac pacing system implantation (i.e. patient implanted with a defibrillator, patient contraindicated for a single dose of 310 μg of dexamethasone sodium phosphate, patient implanted with a tricuspid replacement heart valve, with prior tricuspid valve intervention or with a significant tricuspid valve disease that may lead to future replacement heart valve surgery)
* Minor age patient (i.e. under 18 years of age)
* Incapacitated patient, under guardianship, kept in detention, refusing to cooperate or not able to understand the purpose of this clinical investigation
* Non-menopausal women

Exclusion criteria (phase II):

* Patient planned for a device upgrade, or a device or a lead replacement
* Patient with a congenital heart disease
* Patient with significant hypertrophic cardiomyopathy, cardiac amyloidosis or obstructive hypertrophic cardiomyopathy
* Patient already enrolled in another clinical investigation that could confound the results of this clinical investigation (e.g., clinical investigations involving intra-cardiac device)
* Patient implanted despite a contraindication for cardiac pacing system implantation (i.e. patient implanted with a defibrillator, patient contraindicated for a single dose of 310 μg of dexamethasone sodium phosphate, patient implanted with a tricuspid replacement heart valve, with prior tricuspid valve intervention or with a significant tricuspid valve disease that may lead to future replacement heart valve surgery)
* Minor age patient (i.e. under 18 years of age)
* Incapacitated patient, under guardianship, kept in detention, refusing to cooperate or not able to understand the purpose of this clinical investigation
* Non-menopausal women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-02-14 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Absence of Unanticipated Serious Adverse Device Effect (USADE) related to FLEXIGO delivery catheter | 72 hours after implantation
  Any event caused by use of the FLEXIGO delivery catheter or any accessory packaged with the catheter, will be considered as an ADE related to the FLEXIGO delivery catheter. The primary endpoint evaluation will be based on Sponsor assessment of safety events, based on investigational site reporting.

SECONDARY OUTCOMES:
Implantation success rates | During implantation
  - Implantation success rate with FLEXIGO delivery catheter: Proportion of lead successfully implanted at the interventricular septum with use of the FLEXIGO delivery catheter.
  - Left Bundle Branch Area Pacing (LBBAP) implantation success rate with FLEXIGO delivery catheter: Proportion of lead successfully implanted at the interventricular septum with use of the FLEXIGO delivery catheter and fulfilling LBBAP success criteria according to the operator's decision.
  - LBBAP implantation success rate (overall): Proportion of lead successfully implanted at the interventricular septum with use of any material and fulfilling LBBAP success criteria.
Implantation time | During implantation
  Total procedural time and total fluoroscopic time documented per type of cardiac device implanted and per model of catheter used.
Implantation usability | During implantation
  Implantation usability of the FLEXIGO delivery catheter documented through handling scores based on a specific questionnaire addressed to the operator after implantation.
Serious Adverse Device Effect (SADE) rate related to FLEXIGO delivery catheter or the slitter | 72 hours after implantation
  Proportion of SADE related to the FLEXIGO delivery catheter or the slitter.
Left Bundle Branch Area Pacing (LBBAP) implantation success rate per indication (cardiac pacing and CRT) and per ventricular pacing lead model | During implantation
  - LBBAP implantation success rate with FLEXIGO delivery catheter (documented in cardiac pacing and CRT-D populations separately): Proportion of lead successfully implanted at the interventricular septum with use of the FLEXIGO delivery catheter and fulfilling LBBAP success criteria according to the operator's decision.
  - LBBAP implantation success rate (overall, and documented in cardiac pacing and CRT-D populations separately): Proportion of lead successfully implanted at the interventricular septum with use of any material and fulfilling LBBAP success criteria according to the operator's decision.

CONTACTS AND LOCATIONS:
Locations (3):
- ULS de Coimbra, Coimbra, Portugal
- Spain (2):
  - Hospital Universitario Virgen de las Nieves, Granada
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No